CLINICAL TRIAL: NCT06810973
Title: Substance Use and HIV Action for Reentry and Engagement.
Acronym: SHARE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Anne C Spaulding, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008607; R61DA062365 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: HIV
Keywords: Jail Facilities; ART/PrEP
MeSH Terms: interventions — Sulfamethazine

STUDY DESIGN:
Intervention Model Description: During the two-year R61 phase, the investigators will compare the Intervention vs Enhanced Standard of Care. The investigators will work with new criminal legal institutions and conduct interviews among recently released PWH/PHRS to see how transitional needs in new jurisdictions differ from those experienced by those in FCJ. Building relationships in the R61 phase will position the researchers to scale up a larger study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SUCCESS-E (Experimental): Participants with SUD, living with HIV or at high risk for seroconversion, will be placed in strength-based case management, delivered by a case manager and peer navigators, both in jail and in the community, leading to linkage and retention in healthcare and SUD treatment.
  Interventions: Behavioral: SUCCESS-E
- Control Group (Other): Participants not placed in the intervention group will have healthcare services inform them of possible medical homes for HIV/PrEP care and a list of referral sites for follow-up SUD care.
  Interventions: Behavioral: Enhanced Standard of Care
- Key informant interviews (KII) (Other): Jail staff and community members willing to participate in Key Informant Interviews (KIIs)
  Interventions: Behavioral: Key Informant Interviews

INTERVENTIONS:
Behavioral: SUCCESS-E — SUCCESS-E is a previously developed intervention based on the evidence-based Antiretroviral Treatment and Access to Services (ARTAS) intervention, modified for those detained within a jail system. It is a manualized six-session program delivered by a case management team, composed of a professional case manager and paraprofessional peer navigators.
  In Jail Sessions:
  1. Build Trust
  2. Assess Strengths
  3. Explore life on ART
     Post-Release Sessions:
  4. Link with care
  5. Enhance self-efficacy for HIV care/PrEP
  6. Future transitions
  Other Names: Sustained, Unbroken, Connection to Care Entry Services, and Suppression/Stopping of HIV, Enhanced with Peer Navigators
  Arms: SUCCESS-E
Behavioral: Enhanced Standard of Care — A list of referral sites for follow-up SUD care will be shared. This information sharing without strength-based, longitudinal case management will be an enhancement to treatment as usual. Also, information about HIV/PrEP follow-up in the community will be placed around the jail, such as affixed to the nurses' medication carts that they push from housing unit to unit, twice a day when residents are due for prescription medications.
  Arms: Control Group
Behavioral: Key Informant Interviews — Key informant interviews (KII) will be conducted with jail staff and community stakeholders in the R61 phase to examine perceptions, barriers, and facilitators to SUD and HIV/PrEP service and treatment utilization, as well as document the experiences of SUCCESS-E participants from the pilot phase.
  Other Names: KII
  Arms: Key informant interviews (KII)

SUMMARY:
This study will test a behavioral intervention with a case manager/peer navigator team pairing with clients to deliver transition planning services. The interactions help clients recognize and use their strengths. The goal is to see if this approach improves clients' ability to access healthcare and drug treatment after being released from jail.

DETAILED DESCRIPTION:
The goal of this jail-based study is to test an intervention aimed at helping individuals with substance use disorder (SUD) who have HIV or are at high risk of contracting HIV maintain medications for managing or preventing HIV when transitioning back to the community. Approximately 75% of individuals in jail have SUD and a subset of this group either has HIV or is at risk of seroconversion. People living with HIV require antiretroviral medications to suppress the virus to non-infectious levels, but these medications are often discontinued during the chaotic period following release from jail. Those at risk of HIV can also take antiretroviral therapy as a preventive measure to lower the risk of seroconversion.

Preliminary data suggest that SUCCESS-E, a strengths-based case management and peer navigation program developed via a pilot grant, can help connect individuals to medical care upon release to ensure continued drug therapy. A manual for delivering SUCCESS-E was previously developed to guide case managers and peer navigators.

In this phase, 100 eligible individuals will be enrolled from the Fulton County Jail (FCJ). Participants will be randomly assigned to one of two groups: SUCCESS-E intervention or controls receiving an enhanced version of the jail's discharge planning services.

Data will be collected through medical chart reviews, baseline and follow-up surveys with participants (each taking less than an hour), and single-visit interviews with approximately 30 stakeholders (jail staff, community advocates, and individuals post-program). These key informant interviews will typically last less than an hour and will be recorded for qualitative analysis. Data will also be collected to estimate the cost of delivering the intervention.

The project will apply implementation science to introduce innovations in case management for transitioning individuals from jail back to the community. The case management intervention will be delivered to individuals with HIV or those at high risk of seroconversion, both in jail and post-release. If proven effective, this strategy could help reduce the incidence of new HIV cases by maintaining viral suppression in individuals with HIV and ensuring that those at risk for HIV seroconversion remain on preventive therapy.

The study will focus on individuals, with or without HIV, who have SUD and are either incarcerated or have been released from jails in Georgia within the past six weeks. Participants will ideally be within one week of their release.

The study aims to address the following questions:

* For people without HIV, how can they access a clinic offering HIV prevention medication (Pre-Exposure Prophylaxis, or PrEP)?
* For people living with HIV, how can they access a clinic to receive their HIV medications (Antiretroviral Therapy, or ART)?
* For everyone, how can they get treatment for Substance Use Disorder (SUD)?

ELIGIBILITY:
Inclusion Criteria for Participants:

* Cis- and transgender men and women
* Able to understand and give informed consent
* Willing to participate in study activities
* People with HIV (PWH) or people at high risk of seroconversion (PHRS)
* History of SUD, defined as a score of 2 or more items in the past year on the Justice Community Opioid Innovation Network (JCOIN) SUD assessment tool
* Resident of study jail and agree to participate in the SUCCESS-E program, or released from study jail within six weeks, and agree to participate in the SUCCESS-E program

Inclusion Criteria for Participants in R61 KIIs:

* Participant who completed the intervention or
* A jail administrator/staff member
* Able to give informed consent
* Willing to participate in study activities

Exclusion Criteria:

* Uncontrolled serious mental illness or moderate to severe intellectual impairment, and/or cognitive impairment (inability to comprehend the informed consent document as assessed by study staff during enrollment)
* Admission to a prison facility (Federal or state)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Linkage to ART | 3 months
  Linkage to ART care for individuals with lived experience of HIV or PrEP for PHRS.
Program Retention | 3 months
  Program Retention at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Spaulding, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Fulton County Jail, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be available for sharing.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after study completion.
Access Criteria: Data will be shared electronically with fellow researchers for secondary data analysis by request.